CLINICAL TRIAL: NCT05162131
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of PB2452 (Bentracimab) With and Without Ticagrelor Pretreatment in Chinese Healthy Volunteers
Brief Title: Study to Evaluate the Safety, Tolerability, PK, and PD of PB2452 With and Without Ticagrelor Pretreatment in Chinese Healthy Volunteers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: After recruitment of Cohorts 1-4 was completed, Sponsor decided to terminate study, initially due to COVID and then considering that PK data from the dose planned to be tested in Cohort 5 (18000 mg) would be available from the ongoing Phase 3 study.
Sponsor: SFJ Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PB2452-PT-CL-0006
Record Dates: First submitted 2021-12-02; First posted 2021-12-17 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Healthy
Keywords: Ticagrelor; Platelet Aggregation Inhibitors; P2Y12 Receptor Antagonists
MeSH Terms: interventions — PB-2452

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- 1-a: 100 mg Bentracimab (PB2452) (no Placebo, no Ticagrelor) (Experimental): PB2452 Infusion
  Interventions: Drug: Bentracimab (PB2452) 100 mg or Placebo
- 1-b: 300 mg Bentracimab (PB2452) (no Placebo, no Ticagrelor) (Experimental): PB2452 Infusion
  Interventions: Drug: Bentracimab (PB2452) 300 mg or Placebo
- 1-c: 1000 mg Bentracimab (PB2452) or Placebo (no Ticagrelor) (Experimental): PB2452 Infusion or Placebo - Sodium Chloride
  Interventions: Drug: Bentracimab (PB2452) 1000 mg or Placebo
- 2: 1000 mg Bentracimab (PB2452) or Placebo (Ticagrelor Pre-treatment) (Experimental): PB2452 Infusion or Placebo - Sodium Chloride with Ticagrelor Oral Tablet: 180 mg + 90 mg bid for a total of 5 doses
  Interventions: Drug: Bentracimab (PB2452) 1000 mg or Placebo (With Ticagrelor Pre-Treatment)
- 3: 3000 mg Bentracimab (PB2452) or Placebo (Ticagrelor Pre-treatment) (Experimental): PB2452 Infusion or Placebo - Sodium Chloride with Ticagrelor Oral Tablet: 180 mg + 90 mg bid for a total of 5 doses
  Interventions: Drug: Bentracimab (PB2452) 3000 mg or Placebo (With Ticagrelor Pre-Treatment)
- 4: 9000 mg Bentracimab (PB2452) or Placebo (Ticagrelor Pre-treatment) (Experimental): PB2452 Infusion or Placebo - Sodium Chloride with Ticagrelor Oral Tablet: 180 mg + 90 mg bid for a total of 5 doses
  Interventions: Drug: Bentracimab (PB2452) 9000 mg or Placebo (With Ticagrelor Pre-Treatment)
- 5: 18000 mg Bentracimab (PB2452) or Placebo (Ticagrelor Pre-treatment) (Experimental): PB2452 Infusion or Placebo - Sodium Chloride with Ticagrelor Oral Tablet: 180 mg + 90 mg bid for a total of 5 doses
  Interventions: Drug: Bentracimab (PB2452) 18000 mg or Placebo (With Ticagrelor Pre-Treatment)

INTERVENTIONS:
Drug: Bentracimab (PB2452) 100 mg or Placebo — Experiment 1-a: 100 mg Bentracimab (PB2452) (no Placebo, no Ticagrelor)
  Drug: PB2452 infusion 30 minute - 12-hour infusion
  Arms: 1-a: 100 mg Bentracimab (PB2452) (no Placebo, no Ticagrelor)
Drug: Bentracimab (PB2452) 300 mg or Placebo — Experiment 1-b: 300 mg Bentracimab (PB2452) (no Placebo, no Ticagrelor)
  Drug: PB2452 infusion 30 minute - 12-hour infusion
  Arms: 1-b: 300 mg Bentracimab (PB2452) (no Placebo, no Ticagrelor)
Drug: Bentracimab (PB2452) 1000 mg or Placebo — Experiment 1-c: 1000 mg Bentracimab (PB2452) or Placebo (no Ticagrelor)
  Drug: PB2452 Infusion 30 minute - 12-hour infusion
  Drug: Placebo - Sodium Chloride 30 minute - 12-hour infusion
  Arms: 1-c: 1000 mg Bentracimab (PB2452) or Placebo (no Ticagrelor)
Drug: Bentracimab (PB2452) 1000 mg or Placebo (With Ticagrelor Pre-Treatment) — Experiment 2: 1000 mg Bentracimab (PB2452) or Placebo (Ticagrelor Pre-treatment)
  Drug: PB2452 infusion 30 minute - 12-hour infusion
  Drug: Placebo - Sodium Chloride 30 minute - 12-hour infusion
  Drug: Ticagrelor Oral Tablet - Pre-treatment Ticagrelor 180 mg + 90 mg bid for 5 doses prior to PB2452 or Placebo
  Arms: 2: 1000 mg Bentracimab (PB2452) or Placebo (Ticagrelor Pre-treatment)
Drug: Bentracimab (PB2452) 3000 mg or Placebo (With Ticagrelor Pre-Treatment) — Experiment 3: 3000 mg Bentracimab (PB2452) or Placebo (Ticagrelor Pre-treatment)
  Drug: PB2452 infusion 30 minute - 12-hour infusion
  Drug: Placebo - Sodium Chloride 30 minute - 12-hour infusion
  Drug: Ticagrelor Oral Tablet - Pre-treatment Ticagrelor 180 mg + 90 mg bid for 5 doses prior to PB2452 or Placebo
  Arms: 3: 3000 mg Bentracimab (PB2452) or Placebo (Ticagrelor Pre-treatment)
Drug: Bentracimab (PB2452) 9000 mg or Placebo (With Ticagrelor Pre-Treatment) — Experiment 4: 9000 mg Bentracimab (PB2452) or Placebo (Ticagrelor Pre-treatment)
  Drug: PB2452 infusion 30 minute - 12-hour infusion
  Drug: Placebo - Sodium Chloride 30 minute - 12-hour infusion
  Drug: Ticagrelor Oral Tablet - Pre-treatment Ticagrelor 180 mg + 90 mg bid for 5 doses prior to PB2452 or Placebo
  Arms: 4: 9000 mg Bentracimab (PB2452) or Placebo (Ticagrelor Pre-treatment)
Drug: Bentracimab (PB2452) 18000 mg or Placebo (With Ticagrelor Pre-Treatment) — Experiment 5: 18000 mg Bentracimab (PB2452) or Placebo (Ticagrelor Pre-treatment)
  Drug: PB2452 infusion 30 minute - 12-hour infusion
  Drug: Placebo - Sodium Chloride 30 minute - 12-hour infusion
  Drug: Ticagrelor Oral Tablet - Pre-treatment Ticagrelor 180 mg + 90 mg bid for 5 doses prior to PB2452 or Placebo
  Arms: 5: 18000 mg Bentracimab (PB2452) or Placebo (Ticagrelor Pre-treatment)

SUMMARY:
This is a Phase 1, randomized, double-blind, placebo-controlled, single ascending dose, sequential group study to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of PB2452 (Bentracimab) with and without ticagrelor pretreatment when administered to Chinese healthy male and female subjects.

Up to 6 dose levels will be evaluated. This study will have 5 cohorts and a total of 40 subjects with 8 healthy subjects per cohort. Cohort 1 will be split into 3 parts, Cohort 1-a, 1-b and 1-c. The starting dose of PB2452 will be 100 mg and the planned doses for subsequent parts or cohorts are 300, 1000, 3000, 9000, and 18000 mg.

DETAILED DESCRIPTION:
The study will consist of a screening period (Days -28 to -4), check-in/pretreatment (Day -3 to -1), an in-house treatment period (Days 1 through 4), and follow-up visits (Days 7 and 28 (+2 days)). Subjects will receive an IV dose of study drug on Day 1.

On Day 1, subjects who meet all of the inclusion criteria and none of the exclusion criteria will be assigned to treatment before dosing. For Cohorts 1-c and 2 to 5, subjects will be randomly assigned to receive PB2452 or placebo in a ratio of 3:1.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is born in China to parents and grandparents of Chinese descent. Have not resided more than 5 years outside of China at the time of consent.
2. The subject is male or female 20 ≤ age ≤ 64.
3. The subject has a body mass index 18 ≤ BMI ≤35 kg/m2 and a weight of ≥45 kg but ≤120 kg, inclusive, at screening.
4. The subject is considered by the investigator to be in good general health as determined by medical history, clinical laboratory test results, vital sign measurements, 12-lead ECG results, and physical examination findings at screening.

   Specific inclusionary laboratory values at screening and check-in require the following:
   * Aspartate aminotransaminase (AST), alanine aminotransaminase (ALT), total serum bilirubin and alkaline phosphatase levels without clinically significant abnormality per investigator's discretion
   * White blood cell (WBC) count, platelet count, hemoglobin level without clinically significant abnormality per investigator's discretion
   * Thyroid stimulating hormone (TSH) level without clinically significant abnormality per investigator's discretion at screening
   * Prothrombin time (PT) and partial thromboplastin time (PTT) level without clinically significant abnormality per investigator's discretion
5. Female subjects of childbearing potential must not be pregnant, lactating, or planning to become pregnant before 3 months after the last dose of study drug, and have a negative serum pregnancy test at screening and check-in. Female subjects of childbearing potential must use 2 effective methods of birth control (hormonal contraceptives [i.e., oral, implantable, patch, or injectable contraceptives, hormone-containing intrauterine device that has been in place for at least 2 months prior to screening] in combination with a barrier method [i.e., condoms, sponge, diaphragm, or cervical cap with spermicidal gels or cream]) from 30 days before study drug administration through the end of the study. Double barrier method of condom and spermicide without hormonal contraceptives, or confirmation of sexual abstinence is acceptable, as well as vasectomy for male subjects or male partners of female subjects. Women are considered not to be of childbearing potential if they have fulfilled one of the following criteria: documentation of irreversible surgical sterilization (i.e., hysterectomy, or bilateral oophorectomy [not tubal ligation]), or postmenopausal (defined as amenorrhea for 12 consecutive months following cessation of all exogenous hormonal treatments, and documented plasma follicle-stimulating hormone level >40 IU/mL, or amenorrhea for 24 consecutive months). Male subjects with partners of childbearing potential must agree to use appropriate and effective measures of contraception (e.g., condom plus diaphragm with spermicide; condom plus spermicide) during the study and for 30 days after the last dose of study drug, and to refrain from donating sperm for at least 7 days prior to the dose of study drug and until at least 90 days following the last dose of study drug.
6. The subject agrees to comply with all protocol requirements.
7. The subject is able to provide written informed consent.

Exclusion Criteria:

1. History of any clinically significant acute or chronic disease or medical disorder
2. History or presence of gastrointestinal, hepatic (with the exception of Gilbert's syndrome), or renal disease or renal insufficiency (i.e., estimated glomerular filtration rate <60 ml/min/1.73m2), or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
3. Specific exclusionary criteria for ECG parameters at screening or check-in are any of the following:

   * Prolonged Fridericia-corrected QT interval (QTcF) >450 milliseconds (msec), shortened QTcF <340 msec, or pause >3 seconds, or family history of long QT syndrome
   * Prolonged PR (PQ) interval >240 msec, intermittent second- or third-degree atrioventricular (AV) block or AV dissociation, or shortened PR interval <120 msec
   * Incomplete, full, or intermittent bundle branch block (QRS <110 msec with normal QRS and T wave morphology is acceptable if there is no evidence of left ventricular hypertrophy
4. Any increased risk of bleeding, including the following:

   * Recent history (within 30 days preceding the first dose of study drug) of gastrointestinal bleeding
   * Any history of severe head trauma, intracranial hemorrhage, intracranial neoplasm, arteriovenous malformation, aneurysm, or proliferative retinopathy
   * Any history of intracranial, intraocular, retroperitoneal, or spinal bleeding
   * Any recent (within 30 days preceding the first dose of study drug) major trauma
   * History of hemorrhagic disorders that may increase the risk of bleeding (e.g., hemophilia, von Willebrand's disease)
   * Receiving chronic treatment with nonsteroidal anti-inflammatory drugs (including aspirin [greater than 100 mg daily]), anticoagulants, or other antiplatelet agents that cannot be discontinued (including clopidogrel, prasugrel, ticlopidine, dipyridamole, or cilostazol).
   * Have taken, within 30 days of screening, any anticoagulants including low molecular-weight heparin, or other antiplatelet agents
   * Have taken non-steroidal anti-inflammatory medications, including aspirin within 14 days of screening
5. The subject has a positive test result for hepatitis B surface antigen, hepatitis C virus antibody, or human immunodeficiency virus types 1 or 2 antibodies at screening.
6. Concomitant oral or IV therapy with strong CYP3A inhibitors, CYP3A substrates with narrow therapeutic indices, or strong CYP3A inducers, which cannot be stopped within at least 5 half-lives, but not shorter than 10 days, before randomization.
7. Any prescription or over-the-counter medications (except paracetamol [up to 2 g per day] or as indicated per protocol e.g. for birth control), including herbal or nutritional supplements, within 14 days before the first dose of study drug.
8. The subject has consumed grapefruit or grapefruit juice, Seville orange or Seville orange-containing products (e.g., marmalade), or alcohol-, or xanthine-containing products within 48 hours before dosing with study drug.
9. The subject is participating in any other study within 30 days of the administration of study drug in this study.
10. The subject is taking part in a non-medication study which, in the opinion of the investigator, would interfere with the outcome of the study.
11. The subject has received another new chemical entity (defined as a compound which has not been approved for marketing) or any marketed or investigational biologic agent within 30 days of the administration of study drug in this study or 5 half-lives of the experimental medication, whichever is longer.
12. The subject has involvement with any sponsor or study site employee or their close relatives (e.g., spouse, parents, siblings, or children whether biological or legally adopted).
13. The subject has previously received PB2452 or had been randomized to receive study drug in an earlier cohort for this study.
14. The subject is a smoker or has used nicotine or nicotine-containing products (e.g., snuff, nicotine patch, nicotine chewing gum, e- cigarettes, mock cigarettes, or inhalers) within 3 months before the infusion of study drug.
15. The subject has a known or suspected history of alcohol/drug abuse or has a positive test result for drugs of abuse, alcohol, or cotinine at screening or check-in.
16. The subject has been involved in strenuous activity or contact sports within 48 hours before the admission and while confined in the clinical site.
17. The subject has donated blood or plasma within 1 month of screening or any blood donation/loss more than 500 mL during the 3 months prior to the infusion of study drug.
18. The subject has a history of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the investigator or history of hypersensitivity to drugs with a similar chemical structure or class to ticagrelor, any biologic therapeutic agent, or any significant food allergy that could preclude a standard diet in the clinical site.
19. Concern for the inability of the subject to comply with study procedures and/or follow-up, or, in the opinion of the investigator, the subject is not suitable for entry into the study.

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2021-12-25 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of AEs | Time Frame: 60 days - Starting up to 28 days prior to dosing
Incidence of Clinical Laboratory Abnormalities | 30 Day - Starting day of dosing
Vital Sign Measurements - Changes in Diastolic Blood Pressure | 60 days - Starting up to 28 days prior to dosing
Vital Sign Measurements - Changes in Systolic Blood Pressure | 60 days - Starting up to 28 days prior to dosing
Vital Sign Measurements - Changes in Axillary Temperature | 60 days - Starting up to 28 days prior to dosing
Vital Sign Measurements - Changes in Respiratory Rate | 60 days - Starting up to 28 days prior to dosing
Vital Sign Measurements - Changes in Heart Rate | 60 days - Starting up to 28 days prior to dosing
12-Lead ECG - Incidence of clinically significant findings | 60 days - Starting up to 28 days prior to dosing
Cardiac Telemetry Monitoring - Incidence of clinically significant findings | 3 Days - Starting day 1 day prior to dosing up to 2 days after dosing
Physical examination - Incidence of clinically significant findings | 3 Days - Starting day 1 day prior to dosing up to 2 days after dosing
Immunogenicity | 60 days
  Incidence of Immunogenicity

SECONDARY OUTCOMES:
PB2452 Pharmacokinetic profile - (AUC) (Cohort 1-4) | -10 minutes,0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours and 7 days
  Area under the plasma concentration versus time curve (AUC)
PB2452 Pharmacokinetic profile - (AUC) (Cohort 5) | -10 minutes,10 minutes, 30 minutes, 1, 2, 4, 8, 12, 16, 18, 20, 24, 28, 32, 36, 48, 72 hours and 7 days
  Area under the plasma concentration versus time curve (AUC)
PB2452 Pharmacokinetic profile - (AUC0-t) (Cohort 1-4) | -10 minutes,0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours and 7 days
  Area under the plasma concentration versus time curve from time 0 to the time of the last quantifiable concentration (AUC0-t)
PB2452 Pharmacokinetic profile - (AUC0-t) (Cohort 5) | -10 minutes,10 minutes, 30 minutes, 1, 2, 4, 8, 12, 16, 18, 20, 24, 28, 32, 36, 48, 72 hours and 7 days
  Area under the plasma concentration versus time curve from time 0 to the time of the last quantifiable concentration (AUC0-t)
PB2452 Pharmacokinetic profile - Cmax (Cohorts 1-4) | -10 minutes,0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours and 7 days
  Observed maximum plasma concentration
PB2452 Pharmacokinetic profile - Cmax (Cohort 5) | -10 minutes,10 minutes, 30 minutes, 1, 2, 4, 8, 12, 16, 18, 20, 24, 28, 32, 36, 48, 72 hours and 7 days
  Observed maximum plasma concentration
PB2452 Pharmacokinetic profile - Tmax (Cohorts 1-4) | -10 minutes,0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours and 7 days
  Time to reach the observed maximum plasma concentration
PB2452 Pharmacokinetic profile - Tmax (Cohort 5) | -10 minutes,10 minutes, 30 minutes, 1, 2, 4, 8, 12, 16, 18, 20, 24, 28, 32, 36, 48, 72 hours and 7 days
  Time to reach the observed maximum plasma concentration
PB2452 Pharmacokinetic profile - AUC(0-inf) (Cohorts 1-4) | -10 minutes,0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours and 7 days
  AUC from time 0 extrapolated to infinity
PB2452 Pharmacokinetic profile - AUC(0-inf) (Cohort 5) | -10 minutes, 10 minutes, 30 minutes, 1, 2, 4, 8, 12, 16, 18, 20, 24, 28, 32, 36, 48, 72 hours and 7 days
  AUC from time 0 extrapolated to infinity
PB2452 Pharmacokinetic profile - t½ (Cohorts 1-4) | -10 minutes,0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours and 7 days
  Terminal elimination half-life
PB2452 Pharmacokinetic profile - t½ (Cohort 5) | -10 minutes,10 minutes, 30 minutes, 1, 2, 4, 8, 12, 16, 18, 20, 24, 28, 32, 36, 48, 72 hours and 7 days
  Terminal elimination half-life
PB2452 Pharmacokinetic profile - CL (Cohorts 1-4) | -10 minutes,0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours and 7 days
  Apparent clearance
PB2452 Pharmacokinetic profile - CL (Cohort 5) | -10 minutes,10 minutes, 30 minutes, 1, 2, 4, 8, 12, 16, 18, 20, 24, 28, 32, 36, 48, 72 hours and 7 days
  Apparent clearance
Ticagrelor and Ticagrelor Active Metabolite (TAM) Pharmacokinetic profile - Cmax (Cohorts 2-4) | -10 minutes,0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 hours
  Observed maximum plasma concentration
Ticagrelor and Ticagrelor Active Metabolite (TAM) Pharmacokinetic profile - Cmax (Cohort 5) | -10 minutes,10 minutes, 30 minutes, 1, 2, 4, 8, 12, 16, 18, 20, 24, 28, 32, 36, 48 hours
  Observed maximum plasma concentration
Ticagrelor and Ticagrelor Active Metabolite (TAM) Pharmacokinetic profile - Tmax (Cohorts 2-4) | -10 minutes,0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 hours
  Time to reach the observed maximum plasma concentration
Ticagrelor and Ticagrelor Active Metabolite (TAM) Pharmacokinetic profile - Tmax (Cohort 5) | -10 minutes,10 minutes, 30 minutes, 1, 2, 4, 8, 12, 16, 18, 20, 24, 28, 32, 36, 48 hours
  Time to reach the observed maximum plasma concentration
Ticagrelor and Ticagrelor Active Metabolite (TAM) Pharmacokinetic profile - AUC(0-12) (Cohorts 2-4) | -10 minutes,0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 hours
  AUC from time 0 to 12 hours after dosing
Ticagrelor and Ticagrelor Active Metabolite (TAM) Pharmacokinetic profile - AUC(0-12) (Cohort 5) | -10 minutes,10 minutes, 30 minutes, 1, 2, 4, 8, 12, 16, 18, 20, 24, 28, 32, 36, 48 hours
  AUC from time 0 to 12 hours after dosing
Ticagrelor and Ticagrelor Active Metabolite (TAM) Pharmacokinetic profile - AUC(0-24) (Cohorts 2-4) | -10 minutes,0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 hours
  AUC from time 0 to 24 hours after dosing
Ticagrelor and Ticagrelor Active Metabolite (TAM) Pharmacokinetic profile - AUC(0-24) (Cohort 5) | -10 minutes,10 minutes, 30 minutes, 1, 2, 4, 8, 12, 16, 18, 20, 24, 28, 32, 36, 48 hours
  AUC from time 0 to 24 hours after dosing
Ticagrelor and Ticagrelor Active Metabolite (TAM) Pharmacokinetic profile - AUC(0-48) (Cohorts 2-4) | -10 minutes,0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 hours
  AUC from time 0 to 48 hours after dosing
Ticagrelor and Ticagrelor Active Metabolite (TAM) Pharmacokinetic profile - AUC(0-48) (Cohort 5) | -10 minutes,10 minutes, 30 minutes, 1, 2, 4, 8, 12, 16, 18, 20, 24, 28, 32, 36, 48 hours
  AUC from time 0 to 48 hours after dosing
Ticagrelor and Ticagrelor Active Metabolite (TAM) Pharmacokinetic profile - (Clast) AUC(0-t) (Cohorts 2-4) | -10 minutes,0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 hours
  AUC from time 0 to the time of last quantifiable concentration
Ticagrelor and Ticagrelor Active Metabolite (TAM) Pharmacokinetic profile - (Clast) AUC(0-t) (Cohort 5) | -10 minutes,10 minutes, 30 minutes, 1, 2, 4, 8, 12, 16, 18, 20, 24, 28, 32, 36, 48 hours
  AUC from time 0 to the time of last quantifiable concentration
Ticagrelor and Ticagrelor Active Metabolite (TAM) Pharmacokinetic profile - AUC0-inf (Cohorts 2-4) | -10 minutes,0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 hours
  AUC from time 0 extrapolated to infinity
Ticagrelor and Ticagrelor Active Metabolite (TAM) Pharmacokinetic profile - AUC0-inf (Cohort 5) | -10 minutes,10 minutes, 30 minutes, 1, 2, 4, 8, 12, 16, 18, 20, 24, 28, 32, 36, 48 hours
  AUC from time 0 extrapolated to infinity
Ticagrelor and Ticagrelor Active Metabolite (TAM) Pharmacokinetic profile - t½ (Cohorts 2-4) | -10 minutes,0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 hours
  Terminal elimination half-life (if data permit)
Ticagrelor and Ticagrelor Active Metabolite (TAM) Pharmacokinetic profile - t½ (Cohort 5) | -10 minutes,10 minutes, 30 minutes, 1, 2, 4, 8, 12, 16, 18, 20, 24, 28, 32, 36, 48 hours
  Terminal elimination half-life
Urine Pharmacokinetic profile - Ae24 (Cohorts 1-5) | Before dosing (Pre-dose) and 0 to 6, 6 to 12, 12 to 24 hours, and 24 to 48 hours after the initiation of the study drug infusion
  Total amount of drug excreted in urine at 24 hours after dosing
Urine Pharmacokinetic profile - Ae48 (Cohorts 1-5) | Before dosing (Pre-dose) and 0 to 6, 6 to 12 , 12 to 24, and 24 to 48 hours after the initiation of the study drug infusion
  Total amount of drug excreted in urine at 48 hours after dosing
Urine Pharmacokinetic profile - (Ae t1 - t2 hours) (Cohorts 1-5) | 0 to 6 hours, 6 to 12 hours, 12 to 24 and 24 to 48 hours after the initiation of the study drug infusion
  Total amount of drug excreted in urine at 48 hours after dosing
Urine Pharmacokinetic profile - Fe24 (Cohorts 1-5) | 1 to 24 hours after dosing
  Fraction excreted in urine
Urine Pharmacokinetic profile - Fe48 (Cohorts 1-5) | 1 to 48 hours after dosing
  Fraction excreted in urine
Urine Pharmacokinetic profile - Renal clearance (CLr) for 24 hours (Cohorts 1-5) | 24 hours after dosing
  Renal clearance
Urine Pharmacokinetic profile - Renal clearance (CLr) for 48 hours (Cohorts 1-5) | 48 hours after dosing
  Renal clearance
Ticagrelor and Ticagrelor Active Metabolite (TAM) Urine Pharmacokinetic profile - Ae24 (Cohorts 2-5) | 24 hours after dosing
  Total amount of drug excreted in urine
Ticagrelor and Ticagrelor Active Metabolite (TAM) Urine Pharmacokinetic profile - Ae48 (Cohorts 2-5) | 48 hours after dosing
  Total amount of drug excreted in urine
Ticagrelor and Ticagrelor Active Metabolite (TAM) Urine Pharmacokinetic profile - Aet1-t2 (Cohorts 2-5) | 0 to 6, 6 to 12,12 to 24 and 24 to 48 hours
  Ae from time t1 to t2 hours
Ticagrelor and Ticagrelor Active Metabolite (TAM) Urine Pharmacokinetic profile - Fe24 (Cohorts 2-5) | 1 to 24 hours after dosing
  Fraction excreted in urine
Ticagrelor and Ticagrelor Active Metabolite (TAM) Urine Pharmacokinetic profile - Fe48 (Cohorts 2-5) | 1 to 48 hours after dosing
  Fraction excreted in urine
Ticagrelor and Ticagrelor Active Metabolite (TAM) Urine Pharmacokinetic profile - Renal clearance (CLr) for 24 hours (Cohorts 2-5) | 24 hours after dosing
  Renal clearance
Ticagrelor and Ticagrelor Active Metabolite (TAM) Urine Pharmacokinetic profile - Renal clearance (CLr) for 48 hours (Cohorts 2-5) | 48 hours after dosing
  Renal clearance
Effectiveness of single ascending doses of PB2452 - PRU at each assessment point - P2Y12 Reaction Units with VerifyNow™ PRUTest™ (Cohorts 2-4) | Day -2 (60 minutes prior to first ticagrelor dose) and Day 1 (-10 minutes, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 and 48 hours)
Effectiveness of single ascending doses of PB2452 - PRU at each assessment point - P2Y12 Reaction Units with VerifyNow™ PRUTest™ (Cohort 5) | Day -2 (60 minutes prior to first ticagrelor dose) and Day 1 (-10 minutes, 10 minutes, 30 minutes, 1, 2, 4, 8, 12, 16, 18, 20, 24, 28, 32, 36 and 48 hours)
Effectiveness of single ascending doses of PB2452 - Percent of baseline in PRU - P2Y12 Reaction Units with VerifyNow™ PRUTest™ (Cohorts 2-4) | Day -2 (60 minutes prior to first ticagrelor dose) and Day 1 (-10 minutes, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 and 48 hours)
Percent of baseline in PRU - P2Y12 Reaction Units with VerifyNow™ PRUTest™ (Cohort 5) | Day -2 (60 minutes prior to first ticagrelor dose) and Day 1 (-10 minutes, 10 minutes, 30 minutes, 1, 2, 4, 8, 12, 16, 18, 20, 24, 28, 32, 36 and 48 hours)
  Effectiveness of single ascending doses of PB2452 -
Maximal PRU - P2Y12 Reaction Units with VerifyNow™ PRUTest™ (Cohorts 2-4) | Day -2 (60 minutes prior to first ticagrelor dose) and Day 1 (-10 minutes, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 and 48 hours)
  Effectiveness of single ascending doses of PB2452
Maximal PRU - P2Y12 Reaction Units with VerifyNow™ PRUTest™ (Cohort 5) | Day -2 (60 minutes prior to first ticagrelor dose) and Day 1 (-10 minutes, 10 minutes, 30 minutes, 1, 2, 4, 8, 12, 16, 18, 20, 24, 28, 32, 36 and 48 hours)
  Effectiveness of single ascending doses of PB2452
Time to maximal PRU - P2Y12 Reaction Units with VerifyNow™ PRUTest™ (Cohorts 2-4) | Day -2 (60 minutes prior to first ticagrelor dose) and Day 1 (-10 minutes, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 and 48 hours)
  Effectiveness of single ascending doses of PB2452
Time to maximal PRU - P2Y12 Reaction Units with VerifyNow™ PRUTest™ (Cohort 5) | Day -2 (60 minutes prior to first ticagrelor dose) and Day 1 (-10 minutes, 10 minutes, 30 minutes, 1, 2, 4, 8, 12, 16, 18, 20, 24, 28, 32, 36 and 48 hours)
  Effectiveness of single ascending doses of PB2452
Time to 200 or greater PRU - P2Y12 Reaction Units with VerifyNow™ PRUTest™ (Cohorts 2-4) | Day -2 (60 minutes prior to first ticagrelor dose) and Day 1 (-10 minutes, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 and 48 hours)
  Effectiveness of single ascending doses of PB2452 -
Time to 200 or greater PRU - P2Y12 Reaction Units with VerifyNow™ PRUTest™ (Cohort 5) | Day -2 (60 minutes prior to first ticagrelor dose) and Day 1 (-10 minutes, 10 minutes, 30 minutes, 1, 2, 4, 8, 12, 16, 18, 20, 24, 28, 32, 36 and 48 hours)
  Effectiveness of single ascending doses of PB2452
Time to 60% or greater of baseline PRU - P2Y12 Reaction Units with VerifyNow™ PRUTest™ (Cohorts 2-4) | Day -2 (60 minutes prior to first ticagrelor dose) and Day 1 (-10 minutes, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 and 48 hours)
  Effectiveness of single ascending doses of PB2452
Time to 60% or greater of baseline PRU - P2Y12 Reaction Units with VerifyNow™ PRUTest™ (Cohort 5) | Day -2 (60 minutes prior to first ticagrelor dose) and Day 1 (-10 minutes, 10 minutes, 30 minutes, 1, 2, 4, 8, 12, 16, 18, 20, 24, 28, 32, 36 and 48 hours)
  Effectiveness of single ascending doses of PB2452
Time to 80% or greater of baseline PRU - P2Y12 Reaction Units with VerifyNow™ PRUTest™ (Cohorts 2-4) | Day -2 (60 minutes prior to first ticagrelor dose) and Day 1 (-10 minutes, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 and 48 hours)
  Effectiveness of single ascending doses of PB2452
Time to 80% or greater of baseline PRU - P2Y12 Reaction Units with VerifyNow™ PRUTest™ (Cohort 5) | Day -2 (60 minutes prior to first ticagrelor dose) and Day 1 (-10 minutes, 10 minutes, 30 minutes, 1, 2, 4, 8, 12, 16, 18, 20, 24, 28, 32, 36 and 48 hours)
  Effectiveness of single ascending doses of PB2452
Time to 90% or greater of baseline PRU - P2Y12 Reaction Units with VerifyNow™ PRUTest™ (Cohorts 2-4) | Day -2 (60 minutes prior to first ticagrelor dose) and Day 1 (-10 minutes, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 and 48 hours)
  Effectiveness of single ascending doses of PB2452
Time to 90% or greater of baseline PRU - P2Y12 Reaction Units with VerifyNow™ PRUTest™ (Cohort 5) | Day -2 (60 minutes prior to first ticagrelor dose) and Day 1 (-10 minutes, 10 minutes, 30 minutes, 1, 2, 4, 8, 12, 16, 18, 20, 24, 28, 32, 36 and 48 hours)
  Effectiveness of single ascending doses of PB2452
PRI at each assessment point - Vasodilator stimulated response by ELISA (Cohorts 2-4) | Day -2 (60 minutes prior to first ticagrelor dose) and Day 1 (-10 minutes, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 and 48 hours)
  Effectiveness of single ascending doses of PB2452
PRI at each assessment point - Vasodilator stimulated response (VASP) by ELISA (Cohort 5) | Day -2 (60 minutes prior to first ticagrelor dose) and Day 1 (-10 minutes, 10 minutes, 30 minutes, 1, 2, 4, 8, 12, 16, 18, 20, 24, 28, 32, 36 and 48 hours)
  Effectiveness of single ascending doses of PB2452
Percent of baseline in PRI - Vasodilator stimulated response (VASP) by ELISA (Cohorts 2-4) | Day -2 (60 minutes prior to first ticagrelor dose) and Day 1 (-10 minutes, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 and 48 hours)
  Effectiveness of single ascending doses of PB2452
Percent of baseline in PRI - Vasodilator stimulated response (VASP) by ELISA (Cohort 5) | Day -2 (60 minutes prior to first ticagrelor dose) and Day 1 (-10 minutes, 10 minutes, 30 minutes, 1, 2, 4, 8, 12, 16, 18, 20, 24, 28, 32, 36 and 48 hours)
  Effectiveness of single ascending doses of PB2452
Maximal PRI - Vasodilator stimulated response (VASP) by ELISA (Cohorts 2-4) | Day -2 (60 minutes prior to first ticagrelor dose) and Day 1 (-10 minutes, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 and 48 hours)
  Effectiveness of single ascending doses of PB2452
Maximal PRI - Vasodilator stimulated response (VASP) by ELISA (Cohort 5) | Day -2 (60 minutes prior to first ticagrelor dose) and Day 1 (-10 minutes, 10 minutes, 30 minutes, 1, 2, 4, 8, 12, 16, 18, 20, 24, 28, 32, 36 and 48 hours)
  Effectiveness of single ascending doses of PB2452
Time to maximal PRI - Vasodilator stimulated response (VASP) by ELISA (Cohorts 2-4) | Day -2 (60 minutes prior to first ticagrelor dose) and Day 1 (-10 minutes, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 and 48 hours)
  Effectiveness of single ascending doses of PB2452
Time to maximal PRI - Vasodilator stimulated response (VASP) by ELISA (Cohort 5) | Day -2 (60 minutes prior to first ticagrelor dose) and Day 1 (-10 minutes, 10 minutes, 30 minutes, 1, 2, 4, 8, 12, 16, 18, 20, 24, 28, 32, 36 and 48 hours)
  Effectiveness of single ascending doses of PB2452
Time to 60% or greater of baseline PRI - Vasodilator stimulated response (VASP) by ELISA (Cohorts 2-4) | Day -2 (60 minutes prior to first ticagrelor dose) and Day 1 (-10 minutes, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 and 48 hours)
  Effectiveness of single ascending doses of PB2452
Time to 60% or greater of baseline PRI - Vasodilator stimulated response (VASP) by ELISA (Cohort 5) | Day -2 (60 minutes prior to first ticagrelor dose) and Day 1 (-10 minutes, 10 minutes, 30 minutes, 1, 2, 4, 8, 12, 16, 18, 20, 24, 28, 32, 36 and 48 hours)
  Effectiveness of single ascending doses of PB2452
Time to 80% or greater of baseline PRI - Vasodilator stimulated response (VASP) by ELISA (Cohort 5) | Day -2 (60 minutes prior to first ticagrelor dose) and Day 1 (-10 minutes, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 and 48 hours)
  Effectiveness of single ascending doses of PB2452
Time to 80% or greater of baseline PRI- Vasodilator stimulated response (VASP) by ELISA (Cohort 5) | Day -2 (60 minutes prior to first ticagrelor dose) and Day 1 (-10 minutes, 10 minutes, 30 minutes, 1, 2, 4, 8, 12, 16, 18, 20, 24, 28, 32, 36 and 48 hours)
  Effectiveness of single ascending doses of PB2452
Time to 90% or greater of baseline PRI - Vasodilator stimulated response (VASP) by ELISA (Cohorts 2-4) | Day -2 (60 minutes prior to first ticagrelor dose) and Day 1 (-10 minutes, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 and 48 hours)
  Effectiveness of single ascending doses of PB2452
Time to 90% or greater of baseline PRI - Vasodilator stimulated response (VASP) by ELISA (Cohort 5) | Day -2 (60 minutes prior to first ticagrelor dose) and Day 1 (-10 minutes, 10 minutes, 30 minutes, 1, 2, 4, 8, 12, 16, 18, 20, 24, 28, 32, 36 and 48 hours)
  Effectiveness of single ascending doses of PB2452

CONTACTS AND LOCATIONS:
Overall Officials: Dong Ruihua, Principal Investigator — Beijing Friendship Hospital, 101 Luyuan Est. Rd., Tongzhou District, Beijing, China
Locations (1):
- Beijing Friendship Hospital, Tongzhou, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No